CLINICAL TRIAL: NCT07322276
Title: Effects of Exercise Timing and Physical Activity Level on Sleep Quality and Body Temperature
Brief Title: Effects of Exercise Timing on Sleep Quality
Acronym: SLEEPCORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 25CH122; 2025-A00957-42 (Other: ANSM)
Record Dates: First submitted 2025-11-21; First posted 2026-01-07 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Healthy Endurance Athlet; Inactive People
Keywords: endurance athletes; exercise timing; sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a single-center, open-label, randomized controlled trial with two parallel crossover groups:
  * "Active" group
  * "Inactive-sedentary" group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Inactive-sedentary" group (Active Comparator): inactive participants that realize 3 experimental conditions: evening exercise, morning exercise and control (no-exercise).
  Interventions: Other: Aerobic Exercise
- "Active" group (Experimental): endurance athletes that realize 3 experimental conditions: evening exercise, morning exercise and control (no-exercise).
  Interventions: Other: Aerobic Exercise

INTERVENTIONS:
Other: Aerobic Exercise — The physical exercise consist of treadmill running at 65% of the maximal aerobic speed (MAP) until exhaustion (time to exhaustion exercise type).

SUMMARY:
Modern lifestyles are marked by a prevalence of sedentary behaviors and physical inactivity, which have been linked to numerous adverse health effects. While regular physical exercise is a well-established countermeasure, exercising in the late afternoon may paradoxically disrupt deep sleep due to increased core body temperature. Inactive and sedentary individuals, who often have impaired autonomic function compared to endurance-trained athletes, may be particularly susceptible to these negative effects, potentially resulting in compromised thermoregulation and exacerbated disruptions to deep sleep, a critical stage of sleep essential for overall recovery. Therefore, this study aims to investigate the impact of aerobic exercise performed in the late afternoon versus morning on: 1) deep sleep and sleep onset latency; and 2) core body temperature and its autonomic regulatory mechanisms on endurance-trained and inactive-sedentary people.

ELIGIBILITY:
Inclusion Criteria:

* Group "Inactive" :No regular exercise practice (inactive people that don't follow the WHO recommendations) and have sedentary behaviors
* Group "Active": Regular exercise (athletes that are specialized in aerobic exercise, with more than 300 minutes per-week over 6 months and practice at regional level).

Exclusion Criteria:

* Have sleep disorders medically diagnosed or detected by sleep forms cutoffs (clinical insomnia by ISI, severe risk of obstructive sleep apnea by Stop-Bang, bad sleep quality by PSQI.
* Have a diagnosed mental health condition requiring treatment
* Have renal, respiratory, cardiovascular or neuromuscular disease medically diagnosed.
* Be pregnant or breastfeeding

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-23 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Duration of deep slow-wave sleep | Once weekly for three weeks (day 1, day 7, day 14, day 21)
  Evaluation of the duration of deep slow-wave sleep (N3 stage) quantified by the EEG signal from polysomnography (Nox A1, Resmed®, USA).

SECONDARY OUTCOMES:
Assessment of core temperature | Once weekly for three weeks (Day 1, Day 7, Day 14, Day 21)
  Assessment of core temperature until the end of the sleep period will be measured using gastrointestinal telemetric pills (eCelsius, Bodycap®, France).
Evaluation of autonomic nervous system thermoregulation | Once weekly for three weeks (Day 1, Day 7, Day 14, Day 21)
  Evaluation of autonomic nervous system thermoregulation through time-domain (R-R intervals in ms)
Evaluation of autonomic nervous system thermoregulation | Once weekly for three weeks (Day 1, Day 7, Day 14, Day 21)
  Evaluation of autonomic nervous system thermoregulation through frequency- domain parameters (in Hz)
Complementary sleep evaluation | Once weekly for three weeks (Day 1, Day 7, Day 14, Day 21)
  Complementary sleep evaluation through analysis of duration of N1, N2, and REM stages (in Percentage of Total Sleep Time)
Complementary sleep evaluation | Once weekly for three weeks (Day 1, Day 7, Day 14, Day 21)
  Complementary sleep evaluation through characteristics of slow waves present in N3 (amplitude in microvolts)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ROCHE, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: Undecided
This study is realized only in St-Etienne university Hospital